CLINICAL TRIAL: NCT04131517
Title: An Open-Label, Randomized, Two-Way Crossover Study to Investigate the Potential Pharmacokinetic Interaction of Padsevonil With Oral Contraceptives in Healthy Female Participants
Brief Title: A Study to Test the Interaction of Padsevonil With Oral Contraceptives in Healthy Female Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on available data, UCB has decided to stop development of padsevonil as adjunctive treatment of focal-onset seizures
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UP0035; 2019-002194-54 (EudraCT Number)
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Healthy Female Participants
Keywords: Padsevonil; Contraceptives; Healthy female participants
MeSH Terms: interventions — padsevonil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral contraceptive (Experimental): Participants will receive oral contraceptive in Period 2 of Sequence A and Period 1 of Sequence B of Part 1 and Part 2.
  Interventions: Drug: Microgynon 30®
- Oral contraceptive + padsevonil (Experimental): Participants will receive padsevonil + oral contraceptive in Period 1 of Sequence A and Period 2 of Sequence B of Part 1 and Part 2.
  Interventions: Drug: Padsevonil; Drug: Microgynon 30®

INTERVENTIONS:
Drug: Padsevonil — Study Medication: Padsevonil Dosage formulation: Oral tablets; 400 mg BID (Part 1) and 200 mg BID (Part 2)
  Arms: Oral contraceptive + padsevonil
Drug: Microgynon 30® — Study Medication: Microgynon 30® Dosage formulation: Oral tablets Dose: Ethinyl estradiol 30 µg + levonorgestrel 150 µg

SUMMARY:
The purpose of the study is to investigate the effect of steady-state padsevonil on the pharmacokinetic of a single dose oral contraceptive.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be aged 18 years of age or greater, at the time of signing the informed consent
* Participant must be a premenopausal female with no indication of abnormal or gestational/lactational hypothalamic-pituitary-ovarian function. Menopause will be defined for the purpose of this study as amenorrhea of ≥12 months for which no other reason has been identified
* Participant must not be pregnant or breastfeeding. Participant must agree to use an effective form of contraception (other than hormonal methods) for the duration of the Treatment Period and for at least 90 days (or 5 terminal half-lives) after the last dose of study medication
* Participant must be in good physical and mental health as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Participant must have body weight of at least 45 kg and body mass index within the range 18 to 30 kg/m^2 (inclusive)

Exclusion Criteria:

* Participant has a history of discontinued use of oral contraceptives (OC) for medical reasons
* Participant has any medical reason that would contraindicate the administration of OC (per label)
* Participant has used any of the following within the specified time period prior to first dose of study medication:

  1. Oral contraceptive or oral hormone replacement therapy within prior 30 days
  2. Implanted hormonal contraceptives within prior 6 months
  3. Injectable contraceptives within prior 12 months
  4. Topical controlled-delivery contraceptives within prior 3 months
  5. Hormone-releasing intrauterine devices ('coils') within prior 3 months
* Participant has other relevant gynecological disorders (such as premature ovarian failure or endometriosis)
* Participant has any clinically relevant electrocardiogram (ECG) finding at the Screening Visit or at Baseline (Day -1) that, in the opinion of the Investigator, increases the risks associated with participating in the study. In addition, any study participant with any of the following findings will be excluded:

  1. QT interval corrected for heart rate using Bazett's formula (QTcB) or Fridericia's formula (QTcF) >450 ms in 2 of 3 ECG recordings;
  2. other conduction abnormalities (defined as PR interval ≥220 ms);
  3. irregular rhythms other than sinus arrhythmia or occasional, rare supraventricular or rare ventricular ectopic beats. In case of an out-of-range result, 1 repeat will be allowed. If the result is out-of-range again, the study participant cannot be included

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0035 001, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

REFERENCES:
- [Derived] Chanteux H, MacPherson M, Kramer H, Otoul C, Okagaki T, Rospo C, De Bruyn S, Watling M, Bani M, Sciberras D. Overview of preclinical and clinical studies investigating pharmacokinetics and drug-drug interactions of padsevonil. Expert Opin Drug Metab Toxicol. 2024 Aug;20(8):841-855. doi: 10.1080/17425255.2024.2373108. Epub 2024 Jul 9. PMID 38932723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in October 2019 and concluded in May 2020. No study participants started Part 2 due to the COVID-19 pandemic. Later, the program developing PSL in focal-onset seizures was stopped and the study was terminated.
Pre-assignment Details: Participant flow refers to the Safety Set (SS). No study participants started Part 2 due to the COVID-19 pandemic. Later, the program developing PSL in focal-onset seizures was stopped and the study was terminated.
Groups:
- Part 1 Sequence A: Participants received padsevonil (PSL) tablets 100 milligrams (mg) up-titrated to 400 mg, orally twice daily (bid) from Day 1 to 6 followed by padsevonil 400 mg bid on Day 7 to 14 along with a single dose of oral contraceptive (OC) Microgynon® 30 (ethinylestradiol 30 microgram [mcg] + levonorgestrel 150 mcg) tablet on Day 13 and, then padsevonil down-titrated from 400 mg to 100 mg bid from Day 15 to 19 during first Treatment Period. Participants received a single dose of OC tablet on Day 34 during second Treatment Period. There was a Washout Period of 14 days between the two Treatment Periods.
- Part 1 Sequence B: Participants received a single dose of OC tablet on Day 1 during first Treatment Period. Participants received padsevonil tablets 100 mg up-titrated to 400 mg, bid on Day 18 to 23 followed by padsevonil 400 mg bid on Day 24 to 31 along with a single dose of OC tablet on Day 30 and, then padsevonil down-titrated from 400 mg to 100 mg bid from Day 32 to 36 during second Treatment Period. There was a Washout Period of 14 days between the two Treatment Periods.
Period: Overall Study
Arm/Group | Part 1 Sequence A | Part 1 Sequence B
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to Safety Set which included study participants who received at least 1 dose of study medication (PSL or OC). No study participants started Part 2 due to the COVID-19 pandemic. Later, the program developing PSL in focal-onset seizures was stopped and the study was terminated.
Arm/Group | Part 1 Sequence A | Part 1 Sequence B | Total Title
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (7.3) | 30.0 (9.2) | 35.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 7 | 6 | 13
  Other/Mixed | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ethinylestradiol in Part 1
Description: Cmax is maximum observed plasma concentration of ethinylestradiol (EE). Values were determined from the observed concentration and time data. This outcome measure was planned to be analyzed for 'Oral Contraceptive Alone' and 'PSL + Oral Contraceptive' arms.
Time Frame: Day 13, 14, 15, 34, 35, 36 during Treatment Sequence A and on Day 1, 2, 3, 30, 31 and 32 during Treatment Sequence B
Population: Pharmacokinetic Set (PKS) included all study participants who had no important protocol deviations affecting the PK of EE, LN, or PSL and its metabolite and for whom at least 1 measurable concentration existed.
Measure: Geometric Mean (95% Confidence Interval); unit: picograms per milliliter (pg/mL)
Groups:
- Part 1 Oral Contraceptive Alone (PKS): After OC intake on Day 34 through Day 41 at Sequence A and OC intake on Day 1 through Day 18 (prior to PSL intake) at Sequence B attributed to OC Alone Treatment Period. Participants formed the PKS.
- Part 1 PSL + Oral Contraceptive (PKS): After OC intake on Day 13 with PSL through Day 34 (prior to OC intake) at Sequence A and after OC intake on Day 30 with PSL through Day 43 at Sequence B attributed to PSL + OC Treatment Period. Participants formed the Pharmacokinetic Set (PKS).
Arm/Group | Part 1 Oral Contraceptive Alone (PKS) | Part 1 PSL + Oral Contraceptive (PKS)
Number analyzed (Participants) | 14 | 14
picograms per milliliter (pg/mL) | 41.17 [34.07 to 49.76] | 42.83 [36.23 to 50.65]
Statistical Analysis 1: Comparison: Part 1 Oral Contraceptive Alone (PKS) vs Part 1 PSL + Oral Contraceptive (PKS); The analysis of variance model (ANOVA) included Treatment, Period, and Sequence as fixed effects and participant within Sequence as a random effect; Test type: Other — A lack of PSL effect on EE and LN would have been concluded if the 90% CI of the geometric mean ratio between treatment with PSL + OC and OC Alone of the least squares (LS) means for the log-transformed Cmax was within the bioequivalence acceptance range of 80% to 125%; Geometric LS Mean ratio = 1.0404, 90% CI 2-sided [0.94156 to 1.1497]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Levonorgestrel in Part 1
Description: Cmax is maximum observed plasma concentration of levonorgestrel. Values were determined from the observed concentration and time data. This outcome measure was planned to be analyzed for 'Oral Contraceptive Alone' and 'PSL + Oral Contraceptive' arms.
Time Frame: Day 13, 14, 15, 34, 35, 36 during Treatment Sequence A and on Day 1, 2, 3, 30, 31 and 32 during Treatment Sequence B
Population: Pharmacokinetic Set included all study participants who had no important protocol deviations affecting the PK of EE, LN, or PSL and its metabolite and for whom at least 1 measurable concentration existed.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Part 1 Oral Contraceptive Alone (PKS) | Part 1 PSL + Oral Contraceptive (PKS)
Number analyzed (Participants) | 14 | 14
pg/mL | 2868 [2204 to 3733] | 2560 [2045 to 3206]
Statistical Analysis 1: Comparison: Part 1 Oral Contraceptive Alone (PKS) vs Part 1 PSL + Oral Contraceptive (PKS); The ANOVA model included Treatment, Period, and Sequence as fixed effects and participant within Sequence as a random effect; Test type: Other — A lack of PSL effect on EE and LN would have been concluded if the 90% CI of the geometric mean ratio between treatment with PSL + OC and OC Alone of the LS means for the log-transformed Cmax was within the bioequivalence acceptance range of 80% to 125%; Geometric LS Mean ratio = 0.89272, 90% CI 2-sided [0.76892 to 1.0364]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ethinylestradiol in Part 2
Description: Cmax is maximum observed plasma concentration of ethinylestradiol.
Time Frame: Day 9, 10, 11, 26, 27 and 28 during Treatment Sequence A and on Day 1, 2, 3, 26, 27 and 28 during Treatment Sequence B
Population: Analysis of this outcome measure was not performed because no study participants started Part 2 due to the COVID-19 pandemic. Later, the study was terminated.
Groups:
- Part 2 Oral Contraceptive Alone; Part 2 PSL + Oral Contraceptive: No study participants started Part 2 due to the COVID-19 pandemic. Later, study was terminated.
Arm/Group | Part 2 Oral Contraceptive Alone | Part 2 PSL + Oral Contraceptive
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Levonorgestrel in Part 2
Description: Cmax is maximum observed plasma concentration of levonorgestrel.
Time Frame: Day 9, 10, 11, 26, 27 and 28 during Treatment Sequence A and on Day 1, 2, 3, 26, 27 and 28 during Treatment Sequence B
Population: No study participants started Part 2 due to the COVID-19 pandemic. Later, the program developing PSL in focal-onset seizures was stopped and the study was terminated.
Arm/Group | Part 2 Oral Contraceptive Alone | Part 2 PSL + Oral Contraceptive
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC[0-inf]) of Ethinylestradiol in Part 1
Description: Area under the concentration time curve from time 0 extrapolated to infinity for ethinylestradiol was reported. This outcome measure was planned to be analyzed for 'Oral Contraceptive Alone' and 'PSL + Oral Contraceptive' arms.
Time Frame: Day 13, 14, 15, 34, 35, 36 during Treatment Sequence A and on Day 1, 2, 3, 30, 31 and 32 during Treatment Sequence B
Population: Pharmacokinetic Set included all study participants who had no important protocol deviations affecting the PK of EE, LN, or PSL and its metabolite and for whom at least 1 measurable concentration existed. Here, Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: hours*picograms per milliliter (h*pg/mL)
Arm/Group | Part 1 Oral Contraceptive Alone (PKS) | Part 1 PSL + Oral Contraceptive (PKS)
Number analyzed (Participants) | 13 | 13
hours*picograms per milliliter (h*pg/mL) | 614.6 [513.7 to 735.5] | 629.5 [535.3 to 740.4]
Statistical Analysis 1: Comparison: Part 1 Oral Contraceptive Alone (PKS) vs Part 1 PSL + Oral Contraceptive (PKS); [analysis description as in outcome 2, analysis 1]; Test type: Other — A lack of PSL effect on EE and LN would have been concluded if the 90% CI of the geometric mean ratio between treatment with PSL + OC and OC Alone of the LS means for the log-transformed AUC0-inf was within the bioequivalence acceptance range of 80% to 125%; Geometric LS Mean ratio = 1.0276, 90% CI 2-sided [0.95544 to 1.1052]

6. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC[0-inf]) of Levonorgestrel in Part 1
Description: AUC0-inf is the area under the concentration time curve from time 0 extrapolated to infinity for levonorgestrel was reported. This outcome measure was planned to be analyzed for 'Oral Contraceptive Alone' and 'PSL + Oral Contraceptive' arms.
Time Frame: Day 13, 14, 15, 34, 35, 36 during Treatment Sequence A and on Day 1, 2, 3, 30, 31 and 32 during Treatment Sequence B
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: h*pg/mL
Arm/Group | Part 1 Oral Contraceptive Alone (PKS) | Part 1 PSL + Oral Contraceptive (PKS)
Number analyzed (Participants) | 5 | 8
h*pg/mL | NA [NA to NA] — As pre-specified in the Protocol/Statistical Analysis Plan, Geometric Means, SDs and CVs are only calculated if at least 2/3 of the parameters are properly determined parameters (i.e. calculated and non-flagged). Statistical analysis of ANOVA does not have a data limitation and was pre-specified to be calculated on all available data. | NA [NA to NA] — As pre-specified in the Protocol/Statistical Analysis Plan, Geometric Means, SDs and CVs are only calculated if at least 2/3 of the parameters are properly determined parameters (i.e. calculated and non-flagged). Statistical analysis of ANOVA does not have a data limitation and was pre-specified to be calculated on all available data.
Statistical Analysis 1: Comparison: Part 1 Oral Contraceptive Alone (PKS) vs Part 1 PSL + Oral Contraceptive (PKS); [analysis description as in outcome 2, analysis 1]; Test type: Other — A lack of PSL effect on EE and LN would have been concluded if the 90% CI of the geometric mean ratio between treatment with PSL+ OC and OC Alone of the LS means for the log-transformed AUC0-inf was within the bioequivalence acceptance range of 80% to 125%; Geometric LS Mean ratio = 0.88808, 90% CI 2-sided [0.52185 to 1.5113]

7. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC[0-inf]) of Ethinylestradiol in Part 2
Description: AUC0-inf is the area under the concentration time curve from time 0 extrapolated to infinity of ethinylestradiol.
Time Frame: Day 9, 10, 11, 26, 27 and 28 during Treatment Sequence A and on Day 1, 2, 3, 26, 27 and 28 during Treatment Sequence B
Population: as for outcome 3
Arm/Group | Part 2 Oral Contraceptive Alone | Part 2 PSL + Oral Contraceptive
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC[0-inf]) of Levonorgestrel in Part 2
Description: AUC0-inf is the area under the concentration time curve from time 0 extrapolated to infinity of levonorgestrel.
Time Frame: Day 9, 10, 11, 26, 27 and 28 during Treatment Sequence A and on Day 1, 2, 3, 26, 27 and 28 during Treatment Sequence B
Population: as for outcome 3
Arm/Group | Part 2 Oral Contraceptive Alone | Part 2 PSL + Oral Contraceptive
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) in Part 1
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs were defined as AEs with a start date/time on or after the first dose of study medication (OC or PSL) or any unresolved event already present before administration of study medication that worsened in intensity following exposure to the treatment.
Time Frame: From Baseline up to Safety Follow-Up during Treatment Sequences A and B (up to Day 46)
Population: Safety Set included study participants who received at least 1 dose of study medication (PSL or OC).
Measure: Number; unit: percentage of participants
Groups:
- Part 1 PSL + Oral Contraceptive (SS): After OC intake on Day 13 with PSL through Day 34 (prior to OC intake) at Sequence A and after OC intake on Day 30 with PSL through Day 43 at Sequence B attributed to PSL + OC Treatment Period. Participants formed the Safety Set (SS).
- Part 1 Oral Contraceptive Alone (SS): After OC intake on Day 34 through Day 41 at Sequence A and OC intake on Day 1 through Day 18 (prior to PSL intake) at Sequence B attributed to OC Alone Treatment Period. Participants formed the SS.
- Part 1 PSL Alone (SS): First intake of PSL through Day 13 (prior to OC intake) at Sequence A and PSL intake on Day 18 through Day 30 (prior to OC intake) at Sequence B attributed to PSL Alone Treatment Period. Participants formed the SS.
Arm/Group | Part 1 PSL + Oral Contraceptive (SS) | Part 1 Oral Contraceptive Alone (SS) | Part 1 PSL Alone (SS)
Number analyzed (Participants) | 14 | 14 | 14
percentage of participants | 85.7 | 50.0 | 100.0

10. Secondary Outcome: Percentage of Participants With Serious TEAEs in Part 1
Description: Serious AEs were defined as any untoward medical occurrence that resulted in death, is life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability, is a congenital anomaly, or is an important medical event which based on medical or scientific judgement may jeopardize the participants, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline up to Safety Follow-Up during Treatment Sequences A and B (up to Day 46)
Population: Safety Set included study participants who received at least 1 dose of study medication (PSL or OC).
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 PSL + Oral Contraceptive (SS) | Part 1 Oral Contraceptive Alone (SS) | Part 1 PSL Alone (SS)
Number analyzed (Participants) | 14 | 14 | 14
percentage of participants | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With TEAEs in Part 2
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs were defined as AEs with a start date/time on or after the first dose of study medication (OC or PSL) or any unresolved event already present before administration of study medication that worsened in intensity following exposure to the treatment.
Time Frame: From Baseline up to Safety Follow-Up during Treatment Sequences A and B (up to Day 42)
Population: as for outcome 3
Groups:
- Part 2 PSL Alone: No study participants started Part 2 due to the COVID-19 pandemic. Later, study was terminated.
Arm/Group | Part 2 Oral Contraceptive Alone | Part 2 PSL + Oral Contraceptive | Part 2 PSL Alone
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants With Serious TEAEs in Part 2
Description: as for outcome 10
Time Frame: From Baseline up to Safety Follow-Up during Treatment Sequences A and B (up to Day 42)
Population: as for outcome 3
Arm/Group | Part 2 Oral Contraceptive Alone | Part 2 PSL + Oral Contraceptive | Part 2 PSL Alone
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Steady State Plasma Concentration (Cmax,ss) of Padsevonil in Part 1
Description: Maximum observed plasma concentration of padsevonil at steady-state was reported. This outcome measure was planned to be analyzed for 'PSL + Oral contraceptive' and 'PSL Alone' arms.
Time Frame: Day 12 and 13 (Sequence A) and Day 29 and 30 (Sequence B)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Groups:
- Part 1 PSL Alone (PKS): First intake of PSL through Day 13 (prior to OC intake) at Sequence A and PSL intake on Day 18 through Day 30 (prior to OC intake) at Sequence B attributed to PSL Alone Treatment Period. Participants formed the PKS.
Arm/Group | Part 1 PSL + Oral Contraceptive (PKS) | Part 1 PSL Alone (PKS)
Number analyzed (Participants) | 14 | 14
nanograms per milliliter (ng/mL) | 2008 [1768 to 2281] | 2083 [1899 to 2286]
Statistical Analysis 1: Comparison: Part 1 PSL + Oral Contraceptive (PKS) vs Part 1 PSL Alone (PKS); [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; Geometric LS Mean ratio = 0.96378, 90% CI 2-sided [0.85043 to 1.0922]

14. Secondary Outcome: Steady State Plasma Concentration (Cmax,ss) of Padsevonil in Part 2
Description: Cmax,ss is the steady state plasma concentration of padsevonil.
Time Frame: Day 8 and 9 (Sequence A) and Day 25 and 26 (Sequence B)
Population: as for outcome 3
Arm/Group | Part 2 PSL + Oral Contraceptive | Part 2 PSL Alone
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Time Tau (AUC[0-tau]) of Padsevonil in Part 1
Description: Area under the concentration-time curve over a dosing interval from time 0 to tau for padsevonil was reported. This outcome measure was planned to be analyzed for 'PSL + Oral contraceptive' and 'PSL Alone' arms.
Time Frame: Day 12 and 13 (Sequence A) and Day 29 and 30 (Sequence B)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Part 1 PSL + Oral Contraceptive (PKS) | Part 1 PSL Alone (PKS)
Number analyzed (Participants) | 14 | 14
hours*nanograms per milliliter (h*ng/mL) | 9612 [8273 to 11170] | 9925 [8769 to 11230]
Statistical Analysis 1: Comparison: Part 1 PSL + Oral Contraceptive (PKS) vs Part 1 PSL Alone (PKS); [analysis description as in outcome 2, analysis 1]; Test type: Other — A lack of PSL effect on EE and LN would have been concluded if the 90% CI of the geometric mean ratio between treatment with PSL + OC and OC Alone of the LS means for the log-transformed AUC was within the bioequivalence acceptance range of 80% to 125%; Geometric LS Mean ratio = 0.96842, 90% CI 2-sided [0.91888 to 1.0206]

16. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Time Tau (AUC[0-tau]) of Padsevonil in Part 2
Description: AUC0-tau is area under the concentration-time curve over a dosing interval from time 0 to tau of padsevonil.
Time Frame: Day 8 and 9 (Sequence A) and Day 25 and 26 (Sequence B)
Population: as for outcome 3
Arm/Group | Part 2 PSL + Oral Contraceptive | Part 2 PSL Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to Safety Follow-Up during Treatment Sequences A and B in Part 1 (up to Day 46)
Description: Treatment-emergent AEs were defined as AEs with a start date/time on or after the first dose of study medication (OC or PSL) or any unresolved event already present before administration of study medication that worsened in intensity following exposure to the treatment. No study participants started Part 2 due to the COVID-19 pandemic.
Arm/Group | Part 1 PSL + Oral Contraceptive (SS) | Part 1 Oral Contraceptive Alone (SS) | Part 1 PSL Alone (SS)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 12/14 | 7/14 | 14/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 PSL + Oral Contraceptive (SS) (N=14) | Part 1 Oral Contraceptive Alone (SS) (N=14) | Part 1 PSL Alone (SS) (N=14)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 2 (2) | 0 (0) | 0 (0)
Withdrawal syndrome (General disorders) | 2 (2) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (10) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 9 (10)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 6 (6)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 11 (11)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3)
Behaviour disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Flat affect (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide threat (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 6 (6)
Communication disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated on 22 May 2020 because the program developing padsevonil in focal-onset seizures was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT04131517/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT04131517/SAP_001.pdf